CLINICAL TRIAL: NCT06974175
Title: Effect of Graminex on Infertility Related to Male Accessory Glands Inflammation. Pilot Study
Brief Title: Effect of Graminex on Infertility Related to Male Accessory Glands Inflammation
Acronym: DEPR_1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5878
Record Dates: First submitted 2024-11-21; First posted 2025-05-15 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Male Infertility; Prostatitis
MeSH Terms: conditions — Infertility, Male; Prostatitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Deprox HP (Experimental): Patients with MAGI that will be given Deprox HP therapy
  Interventions: Other: Deprox_HP
- Group 2: PEA+bromelin+horse chestnut extract (Active Comparator): Patients with MAGI that will be given PEA+bromelin+horse chestnut extract
  Interventions: Other: Peacist

INTERVENTIONS:
Other: Deprox_HP — Use of nutraceutic based on a compound of pollen extracts from pollen, mais and timothy
  Arms: Group 1: Deprox HP
Other: Peacist — Use of a nutraceutic based on palmitoilethanolamide + Bromelin + Horse Chestunt extract
  Arms: Group 2: PEA+bromelin+horse chestnut extract

SUMMARY:
Male Accessory Glands Inflammations (MAGI) include inflammatory diseases involving seminal vescicles and the prostate. Patients suffering from them present an impaired fertility because of seminal duct obstruction and alterations of the rheologic and functional parameters of semen, induced by direct microbiological action as well as inflammatory and oxidative damage. Inflammation in seminal plasma can be detected and measured by dosing of inflammatory molecules such as SuPAR and ST2. Treatment of MAGIs include specific antibiotic therapy in addition to use of anti-inflammatory nutraceutics. Deprox HP is a nutraceutic containing GraminexTM, a compound made of pollen extracts of rye, mais and timothy. To investigate its efficacy, we evalued seminal parameters, inflammatory and oxidative molecules in seminal plasma and clinical and ultrasonographic features of male accessory glands before and after 3 months of treatment in 20 patients taking Deprox HP and 20 patients undergoing treatment with palmitoilethanolammide, bromelin and horse chestnut extract.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with a diagnosis of MAGI based on clinical and/or ultrasonographic criteria.

Exclusion Criteria:

* History of cryptorchidism, orchitis, testicular torsion or trauma,
* Hypogonadism,
* Occupational chemical exposure,
* Y chromosome microdeletions, karyotype abnormalities and Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) mutations,
* ultrasound testicular volume <12 mL,
* FSH >8 mUI/L,
* fever or drug use within 3 months prior to the enrollment in this study
* azoospermia.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Modifications of number of spermatozoa | 6 months
  Modifications of the number of spermatozoa in Millions
Modification of sperm motility | 6 months
  Modification of sperm progressive motility in %
Modifications of number of typical forms | 6 months
  Modifications of number of typical forms in %

SECONDARY OUTCOMES:
Modifications of seminal inflammatory parameters | 6 months
  Modifications of seminal inflammatory parameters ST2 and SuPAR, both expressed in ng/mL
Modifications of seminal oxidative parameters | 6 months
  Modifications of reactive oxygen species expressed in mEq

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Milardi, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

REFERENCES:
- [Result] La Vignera S, Condorelli RA, Vicari E, D'Aagata R, Salemi M, Calogero AE. Hyperviscosity of semen in patients with male accessory gland infection:direct measurement with quantitative viscosimeter. Andrologia. 2012 May;44 Suppl 1:556-9. doi: 10.1111/j.1439-0272.2011.01226.x. Epub 2011 Sep 15. PMID 21919943
- [Result] Gopalkrishnan K, Padwal V, Balaiah D. Does seminal fluid viscosity influence sperm chromatin integrity? Arch Androl. 2000 Sep-Oct;45(2):99-103. doi: 10.1080/014850100418783. PMID 11028927
- [Result] Comhaire FH, Mahmoud AM, Depuydt CE, Zalata AA, Christophe AB. Mechanisms and effects of male genital tract infection on sperm quality and fertilizing potential: the andrologist's viewpoint. Hum Reprod Update. 1999 Sep-Oct;5(5):393-8. doi: 10.1093/humupd/5.5.393. PMID 10582779
- [Result] Alvarez JG, Touchstone JC, Blasco L, Storey BT. Spontaneous lipid peroxidation and production of hydrogen peroxide and superoxide in human spermatozoa. Superoxide dismutase as major enzyme protectant against oxygen toxicity. J Androl. 1987 Sep-Oct;8(5):338-48. doi: 10.1002/j.1939-4640.1987.tb00973.x. PMID 2822642
- [Result] Jones R, Mann T, Sherins R. Peroxidative breakdown of phospholipids in human spermatozoa, spermicidal properties of fatty acid peroxides, and protective action of seminal plasma. Fertil Steril. 1979 May;31(5):531-7. doi: 10.1016/s0015-0282(16)43999-3. PMID 446777
- [Result] Jones R, Mann T. Damage to ram spermatozoa by peroxidation of endogenous phospholipids. J Reprod Fertil. 1977 Jul;50(2):261-8. doi: 10.1530/jrf.0.0500261. PMID 881664
- [Result] Autilio C, Morelli R, Milardi D, Grande G, Marana R, Pontecorvi A, Zuppi C, Baroni S. Soluble urokinase-type plasminogen activator receptor as a putative marker of male accessory gland inflammation. Andrology. 2015 Nov;3(6):1054-61. doi: 10.1111/andr.12084. Epub 2015 Sep 18. PMID 26384478
- [Result] Milardi D, Grande G, Autilio C, Mancini F, De Marinis L, Marana R, Zuppi C, Urbani A, Pontecorvi A, Baroni S. Seminal suPAR Levels as Marker of Abacterial Male Accessory Gland Inflammation in Hypogonadism. Protein Pept Lett. 2018;25(5):478-482. doi: 10.2174/0929866525666180418121421. PMID 29667546
- [Result] Schroder K, Tschopp J. The inflammasomes. Cell. 2010 Mar 19;140(6):821-32. doi: 10.1016/j.cell.2010.01.040. PMID 20303873
- [Result] Di Nicuolo F, Specchia M, Trentavizi L, Pontecorvi A, Scambia G, Di Simone N. An Emerging Role of Endometrial Inflammasome in Reproduction: New Therapeutic Approaches. Protein Pept Lett. 2018;25(5):455-462. doi: 10.2174/0929866525666180412160045. PMID 29651937
- [Result] Inan, S. The Potential Role of Nutraceuticals in Inflammation and Oxidative Stress. IntechOpen. 2020.
- [Result] Zhang X, Ibrahim E, de Rivero Vaccari JP, Lotocki G, Aballa TC, Dietrich WD, Keane RW, Lynne CM, Brackett NL. Involvement of the inflammasome in abnormal semen quality of men with spinal cord injury. Fertil Steril. 2013 Jan;99(1):118-124.e2. doi: 10.1016/j.fertnstert.2012.09.004. Epub 2012 Oct 3. PMID 23040525
- [Result] Cui ZW, Xie ZX, Wang BF, Zhong ZH, Chen XY, Sun YH, Sun QF, Yang GY, Bian LG. Carvacrol protects neuroblastoma SH-SY5Y cells against Fe(2+)-induced apoptosis by suppressing activation of MAPK/JNK-NF-kappaB signaling pathway. Acta Pharmacol Sin. 2015 Dec;36(12):1426-36. doi: 10.1038/aps.2015.90. Epub 2015 Nov 23. PMID 26592517